CLINICAL TRIAL: NCT00169052
Title: Rehabilitation and Health Care for Elderly With SMI
Brief Title: Health Care Management and Rehabilitation Skills Training for Treating Serious Mental Illness in Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH062324 (NIH); R01MH062324 (NIH); DSIR 82-SEMS
Record Dates: First submitted 2005-09-11; First posted 2005-09-15 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2001-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Major Depression
Keywords: geriatric,; older; serious mental illness; SMI
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Depressive Disorder, Major

INTERVENTIONS:
Behavioral: Health Care Management and Supported Rehabilitation

SUMMARY:
This study will evaluate the effectiveness of a health management and supported rehabilitation intervention in treating serious mental illnesses in older people.

DETAILED DESCRIPTION:
This randomized, controlled study will evaluate the effectiveness of a health management (HM) and supported rehabilitation (SR) intervention for 180 older persons (age 50+) with serious mental illness. We will address the following specific aims and hypotheses:

Specific Aim 1- To compare the effectiveness of SR/HM to UC in improving independent living skills and health management. We hypothesize that compared to older individuals with SMI receiving UC, individuals receiving SR/HM will have better independent living skills and health management, evidenced by:

1. Better community living skills and better social skills based on performance-based measures and self-reports of functioning, and
2. Better medication management skills based on performance-based and self-report measures and greater use of preventive and routine primary health care (including annual check-ups with a primary care provider and participation in preventive health care).

Specific Aim 2- To compare the effectiveness of SR/HM to UC in decreasing the use of high-cost acute and long-term institution-based services. We hypothesize that compared to older individuals with SMI receiving UC, individuals receiving SR/HM will use fewer high cost services, including emergency room visits, acute hospitalizations, and nursing home care. In addition, the reduced use of high cost institution-based services will be associated with better independent living skills and health management practices resulting from the SR/HM intervention.

We will also evaluate the following secondary, exploratory hypotheses:

1. The SR/HM intervention will be associated with better general health status.
2. The effectiveness of SR/HM in improving living skills and community functioning will be greatest for individuals with low levels of cognitive impairment.

In addition, we will describe outpatient service utilization for SR/HM and UC models within each study site in order to present a more comprehensive account of services used by study participants.

Little is known about how to provide effective rehabilitation and health management services to older persons with serious mental illness (SMI) to decrease the use of high-cost institution-based services. To address this need, we developed a supported rehabilitation and health management (SR/HM) intervention for older persons with SMI that addresses functioning in two areas essential for preventing hospitalizations and long-term institutional care: (1) enhanced independent living skills and (2) improved health management. The supported rehabilitation (SR) component consists of skills training aimed at improving competence in everyday functioning, including community living skills and social skills. The health management (HM) component consists of training in health management skills and health case management by nurses who monitor and facilitate routine preventive and acute health care. Results from a pilot study indicate that SR/HM is effective in improving independent living skills and health management for older persons with SMI.

The aims of this study are to test the effectiveness of the SR/HM intervention in improving the functioning and health care of older persons with SMI and in reducing the use of high cost, acute and long-term institution-based care. The proposed research will compare the SR/HM intervention to usual care (UC) in a randomized, controlled study of 180 individuals age 60 and older with SMI living in the community.

ELIGIBILITY:
Inclusion Criteria:

* age 50+ with schizophrenia,schizoaffective disorder,bipolar disorder, major depression with functional impairment

Exclusion Criteria:

* dementia, life threatening acute medical condition.

Min Age: 50 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2001-09; Study Completion 2006-08

PRIMARY OUTCOMES:
independent living, social and health behavior skills
preventive health care

SECONDARY OUTCOMES:
Acute emergency, hospitalization and long-term institution-based care

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Bartels, MD, Principal Investigator — Dartmouth
Locations (3):
- United States (3):
  - Freedom Trail Clinic, Boston, Massachusetts
  - Massachusetts Mental Health Center, Boston, Massachusetts
  - Community Council of Nashua, Nashua, New Hampshire